CLINICAL TRIAL: NCT02105155
Title: Non-inferiority and Tolerance of Conversion From Prograf® to Advagraf® at D7 Versus D90 After Liver Transplantation
Brief Title: Conversion Prograf® to Advagraf® at D7 Versus D90 After Liver Transplantation
Acronym: Conversion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P 120907; HAO 2012 (Other: Assistance Publique)
Record Dates: First submitted 2014-04-02; First posted 2014-04-07 (Estimated); Last update posted 2017-12-08 (Actual); Status verified 2017-11

CONDITIONS: Immunosuppression After Liver Transplantation
Keywords: Liver transplantation,; Conversion (Prograf® to Advagraf®),; Prograf® ,; Advagraf® ,; acute rejection,; GFR

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conversion at day 7 ± 3 (Experimental): Conversion from Prograf to Advagraf at D7 ± 3
  Interventions: Drug: Conversion at day 7 ± 3 Prograf® to Advagraf®
- Conversion at day 90±5 (Active Comparator): Conversion from Prograf to Advagraf at 90±5
  Interventions: Drug: Conversion at day 90±5 Prograf® to Advagraf®

INTERVENTIONS:
Drug: Conversion at day 7 ± 3 Prograf® to Advagraf® — Conversion from Prograf® (tacrolimus administered twice daily) to Advagraf® (once-daily prolonged-release tacrolimus) at day 7±3
  Arms: Conversion at day 7 ± 3
Drug: Conversion at day 90±5 Prograf® to Advagraf® — Conversion from Prograf® (tacrolimus administered twice daily) to Advagraf® (once-daily prolonged-release tacrolimus) at day 90±5
  Arms: Conversion at day 90±5

SUMMARY:
The best period for the conversion from Prograf (tacrolimus administered twice daily) to Advagraf (once-daily prolonged-release tacrolimus) remains unknown. The aim of this prospective, randomized, multicenter trial is to prove the non-inferiority of the early conversion (at D7) versus the conversion at D90 after liver transplantation. The primary objective will be to evaluate the incidence of a first biopsy-proven acute rejection in the 6 first months, and prove the non-inferiority of the conversion at D7 + / - 3 versus the conversion at D90 + / - 5 (reference group). If non-inferiority is proved, the two strategies will be compared in terms of superiority. 250 patients will be included. Three ancillary studies will be added : a PK study in a subgroup of 40 patients (20 patients per arm), an assay of the calcineurin activity on a subgroup of 40 patients, and a medicoeconomic study in all patients

DETAILED DESCRIPTION:
Rationale :

Conversion from Prograf (tacrolimus administered twice daily) to Advagraf (once-daily prolonged-release tacrolimus) is currently proposed in both stable and de novo liver transplant recipients. However, the early conversion (around D7 after transplantation), during hospitalization, may be difficult due to the more frequent need of dose adjustments under Advagraf than under Prograf, so that there is no consensus on the best period for the conversion. The aim of this prospective, randomized, multicenter trial is to prove the non-inferiority - in terms of efficacy - of the early conversion (at D7) versus the conversion at D90 after liver transplantation.

Primary objective :

To evaluate the incidence of biopsy-proven acute rejection in the 6 first months after liver transplantation, and prove the non-inferiority of the conversion at D7 + / - 3 versus the conversion at D90 + / - 5 (reference group).

Secondary objectives :

Compare the two strategies in terms of:

* Severity of acute rejection (criteres of Banff 97)
* Steroid-resistant acute rejection
* Number of dose adjustments to obtain the target trough level after conversion
* Patient and graft survival Analyse the PK profile of two subgroups (20 patients in each arm) under Advagraf Measure the calcineurin activity in the two groups (in the patients selected for the PK analysis) Evaluate tolerance, with a particular focus on the renal function at 6 months (glomerular filtration rate using MDRD4) and on adverse events.

Primary endpoint:

Percentage of patients with a first episode of biopsy-proven acute rejection.

Methodology :

Multicenter (13 French liver transplant centers), randomized (central randomisation), open study, of non-inferiority, comparing the efficacy at 6 months of two strategies of conversion from Prograf to Advagraf (D7 + / - 3 versus D90 + / - 5), in addition to mycophenolate mofetil and steroids, in liver transplant recipients. If non-inferiority is proved, the two strategies will be compared in terms of superiority. Inclusion of 250 patients (to analyse at least 112 patients in each arm). Calculation of the sample size is based on the following data: Incidence of acute rejection at 6 months = 20% in the 2 groups, Non-inferiority margin = 15%, alpha risk = 2.5%, power = 80%).

Treatments :

* Prograf introduced at 0,1 - 0,2 mg/kg/day
* Mycophenolate mofetil : 1g TD
* Steroids according to the current use in each center Trough blood concentration of tacrolimus will be 8 - 15 ng/mL during the first 3 months, then 5 à 12 ng/mL thereafter.

PK study: For the 40 patients included in the PK study (20 patients per arm), the PK profile (C0, Cmax and AUC) will be established on 9 points : 0 (before Advagraf administration) then at 20min, 40 min, 60 min, 2h, 3h, 4h, 6h, 8h.

* 7 days after conversion in the first group (early conversion)
* 14 + / - 5 days after conversion in the other group (conversion at D90) Calcineurin activity will be assayed on the blood samples used for the trough concentration determination at D5, D7, M1, M3 and M6 and on a baseline sample.

Medicoeconomic study : The costs induced by liver transplantation will be calculated in all the patients included and randomized according to the French recommendations.

ELIGIBILITY:
Inclusion Criteria :

* 18 to 75 years
* First liver transplantation
* No contra-indication to tacrolimus, mycophenolate mofetil or steroids
* Informed consent signed
* French Health Assurance

Exclusion Criteria :

* Combined transplantation
* Severe uncontrolled infection
* Hypersensitivity to tacrolimus or its excipients, to other macrolides, to mycophenolate mofetil or its excipients
* Pregnant or lactating woman, or women of childbearing potential without adequate method of contraception
* Cancer or pasthistory of cancer other than basal or squamous cell carcinoma or hepatocellular carcinoma suitable for liver transplantation
* Patients with renal impairment where GFR is less than 30ml/min
* HIV positivity

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10-17 (Actual)

PRIMARY OUTCOMES:
First episode of acute rejection during the first 6 months | 6 months
  First episode of acute rejection during the first 6 months

SECONDARY OUTCOMES:
Renal function | 6 months
  Glomerular filtration rate using MDRD4
Adverse effects | 6 months
  All side effects
Severity of acute rejection | 6 months
  Histological severity of acute rejection using the Banff 2007 criteria

CONTACTS AND LOCATIONS:
Overall Officials: Yvon Calmus, MD, PhD, Principal Investigator — Assistance Publique
Locations (1):
- Hôpital Pitié Salpêtrière unité médicale de transplantion hépatique, Paris, France

REFERENCES:
- [Derived] Allard M, Puszkiel A, Conti F, Chevillard L, Kamar N, Noe G, White-Koning M, Thomas-Schoemann A, Simon T, Vidal M, Calmus Y, Blanchet B. Pharmacokinetics and Pharmacodynamics of Once-daily Prolonged-release Tacrolimus in Liver Transplant Recipients. Clin Ther. 2019 May;41(5):882-896.e3. doi: 10.1016/j.clinthera.2019.03.006. Epub 2019 Apr 17. PMID 31003735